CLINICAL TRIAL: NCT01919567
Title: Observational Study on the Carcinogenesis of SOX-9 in Oral Cancer, and Chemopreventive Possibility for the Treatment of Oral Cancer Using SOX-9 Inhibitor.
Brief Title: Study on the Carcinogenesis of SOX-9 in Oral Cancer, and Chemopreventive Possibility for the Treatment of Oral Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201012095RC
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-11

CONDITIONS: Carcinogenesis; Oral Cancer
Keywords: SOX-9; Oral cancer; arecoline
MeSH Terms: conditions — Carcinogenesis; Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — tissue, serum, saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Normal team: Subjects who have problem at third molar of impacted tooth need to receive a surgery with general anesthesia.
  Subjects must:
  Should have a blood exam (20ml) before the surgery.
  Site staff must:
  Collect subjects' saliva once a day (in the morning before breakfast) for 3 consecutive days.
  Collect a 0.5x0.5Cm2 tissue sample around third molar during the surgery.
- Oral dysplasia: Subjects who are diagnosed with dysplasia of oral cavity.
  Subjects must:
  Should have a blood exam (20ml/each time) before the surgery and 3 months after the surgery.
  In the case the disease recurs after the surgery, subjects need to receive the surgery again and take another blood exam before the surgery and 3 months after the surgery.
  Before the surgery site staff must:
  Collect saliva once a day (in the morning before breakfast) for 3 consecutive days.
  Collect a 0.5x0.5Cm2 tissue sample of the tumor during the surgery.
- Oral cancer: Subjects who suffer from oral cancer.
  Subjects must:
  Should have a blood exam (20ml/each time) before the surgery and 3 months after the surgery.
  In the case the disease recurs after the surgery, subjects need to receive the surgery again and take another blood exam before the surgery and 3 months after the surgery.
  Before the surgery site staff must:
  Collect subjects' saliva once a day (in the morning before breakfast) for 3 consecutive days.
  Collect a 0.5x0.5Cm2 tissue sample of the tumor during the surgery.

SUMMARY:
Study on the Carcinogenesis of SOX-9 in Oral Cancer, and Chemopreventive Possibility for the Treatment of Oral Cancer Using SOX-9 Inhibitor.

DETAILED DESCRIPTION:
To find out if there is prognostic value which to the performance of SOX-9 of oral cancer in Taiwan and provide some reference for future treatment.

We anticipate to enroll 40 persons with normal oral mucosa, 65 persons with oral dysplasia and 150 persons with oral cancer and collect the tissue which was stained for pathological sections over a 3 year period.

We also collect the blood and saliva samples from patients and the results along with patient-specific information such as tumor phases, tumor size, lymph node metastasis, cancer metastasis, prognosis and betel nut chewing, smoking and drinking habits and other parameters are statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Dysplasia or cancer of the oral cavity.

Exclusion Criteria:

* pregnant woman

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical center
Sampling Method: Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Carcinogenesis of SOX-9 | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shin-Jung Cheng, DDS, MS, PhD, Principal Investigator
Locations (1):
- National Taiwan University Hospital research Ethics Committee, Taipei, Taiwan

REFERENCES:
- [Background] Afonja O, Raaka BM, Huang A, Das S, Zhao X, Helmer E, Juste D, Samuels HH. RAR agonists stimulate SOX9 gene expression in breast cancer cell lines: evidence for a role in retinoid-mediated growth inhibition. Oncogene. 2002 Nov 7;21(51):7850-60. doi: 10.1038/sj.onc.1205985. PMID 12420222
- [Background] Aleman A, Adrien L, Lopez-Serra L, Cordon-Cardo C, Esteller M, Belbin TJ, Sanchez-Carbayo M. Identification of DNA hypermethylation of SOX9 in association with bladder cancer progression using CpG microarrays. Br J Cancer. 2008 Jan 29;98(2):466-73. doi: 10.1038/sj.bjc.6604143. Epub 2007 Dec 18. PMID 18087279
- [Background] Alvarez-Medina R, Le Dreau G, Ros M, Marti E. Hedgehog activation is required upstream of Wnt signalling to control neural progenitor proliferation. Development. 2009 Oct;136(19):3301-9. doi: 10.1242/dev.041772. PMID 19736325
- [Background] Bien-Willner GA, Stankiewicz P, Lupski JR. SOX9cre1, a cis-acting regulatory element located 1.1 Mb upstream of SOX9, mediates its enhancement through the SHH pathway. Hum Mol Genet. 2007 May 15;16(10):1143-56. doi: 10.1093/hmg/ddm061. Epub 2007 Apr 4. PMID 17409199
- [Background] Lu B, Fang Y, Xu J, Wang L, Xu F, Xu E, Huang Q, Lai M. Analysis of SOX9 expression in colorectal cancer. Am J Clin Pathol. 2008 Dec;130(6):897-904. doi: 10.1309/AJCPW1W8GJBQGCNI. PMID 19019766
- [Background] Drivdahl R, Haugk KH, Sprenger CC, Nelson PS, Tennant MK, Plymate SR. Suppression of growth and tumorigenicity in the prostate tumor cell line M12 by overexpression of the transcription factor SOX9. Oncogene. 2004 Jun 3;23(26):4584-93. doi: 10.1038/sj.onc.1207603. PMID 15077158
- [Background] Wang H, Leav I, Ibaragi S, Wegner M, Hu GF, Lu ML, Balk SP, Yuan X. SOX9 is expressed in human fetal prostate epithelium and enhances prostate cancer invasion. Cancer Res. 2008 Mar 15;68(6):1625-30. doi: 10.1158/0008-5472.CAN-07-5915. PMID 18339840
- [Background] Jay P, Berta P, Blache P. Expression of the carcinoembryonic antigen gene is inhibited by SOX9 in human colon carcinoma cells. Cancer Res. 2005 Mar 15;65(6):2193-8. doi: 10.1158/0008-5472.CAN-04-1484. PMID 15781631
- [Background] Knower KC, Kelly S, Harley VR. Turning on the male--SRY, SOX9 and sex determination in mammals. Cytogenet Genome Res. 2003;101(3-4):185-98. doi: 10.1159/000074336. PMID 14684982
- [Background] Ishida K, Ito S, Wada N, Deguchi H, Hata T, Hosoda M, Nohno T. Nuclear localization of beta-catenin involved in precancerous change in oral leukoplakia. Mol Cancer. 2007 Oct 9;6:62. doi: 10.1186/1476-4598-6-62. PMID 17922924
- [Background] Mertin S, McDowall SG, Harley VR. The DNA-binding specificity of SOX9 and other SOX proteins. Nucleic Acids Res. 1999 Mar 1;27(5):1359-64. doi: 10.1093/nar/27.5.1359. PMID 9973626
- [Background] Murata M, Iwao K, Miyoshi Y, Nagasawa Y, Yabu M, Himeno S, Imanishi K, Ohsawa M, Wada H, Tominaga S, Shimano T, Kobayashi T, Nakamura Y. Activation of the beta-catenin gene by interstitial deletions involving exon 3 as an early event in colorectal tumorigenesis. Cancer Lett. 2000 Oct 16;159(1):73-8. doi: 10.1016/s0304-3835(00)00533-4. PMID 10974408
- [Background] Fracalossi AC, Silva Mde S, Oshima CT, Ribeiro DA. Wnt/beta-catenin signalling pathway following rat tongue carcinogenesis induced by 4-nitroquinoline 1-oxide. Exp Mol Pathol. 2010 Feb;88(1):176-83. doi: 10.1016/j.yexmp.2009.11.004. Epub 2009 Nov 17. PMID 19931241
- [Background] de Camargo Cancela M, Voti L, Guerra-Yi M, Chapuis F, Mazuir M, Curado MP. Oral cavity cancer in developed and in developing countries: population-based incidence. Head Neck. 2010 Mar;32(3):357-67. doi: 10.1002/hed.21193. PMID 19644932
- [Background] Blache P, van de Wetering M, Duluc I, Domon C, Berta P, Freund JN, Clevers H, Jay P. SOX9 is an intestine crypt transcription factor, is regulated by the Wnt pathway, and represses the CDX2 and MUC2 genes. J Cell Biol. 2004 Jul 5;166(1):37-47. doi: 10.1083/jcb.200311021. PMID 15240568
- [Background] Scully C, Bagan J. Oral squamous cell carcinoma overview. Oral Oncol. 2009 Apr-May;45(4-5):301-8. doi: 10.1016/j.oraloncology.2009.01.004. Epub 2009 Feb 26. No abstract available. PMID 19249237
- [Background] Supic G, Kozomara R, Brankovic-Magic M, Jovic N, Magic Z. Gene hypermethylation in tumor tissue of advanced oral squamous cell carcinoma patients. Oral Oncol. 2009 Dec;45(12):1051-7. doi: 10.1016/j.oraloncology.2009.07.007. Epub 2009 Aug 8. PMID 19665921
- [Background] Vidal VP, Ortonne N, Schedl A. SOX9 expression is a general marker of basal cell carcinoma and adnexal-related neoplasms. J Cutan Pathol. 2008 Apr;35(4):373-9. doi: 10.1111/j.1600-0560.2007.00815.x. PMID 18333897
- [Background] Koopman P, Bullejos M, Bowles J. Regulation of male sexual development by Sry and Sox9. J Exp Zool. 2001 Sep 15;290(5):463-74. doi: 10.1002/jez.1089. PMID 11555853
- [Background] Jiang SS, Fang WT, Hou YH, Huang SF, Yen BL, Chang JL, Li SM, Liu HP, Liu YL, Huang CT, Li YW, Jang TH, Chan SH, Yang SJ, Hsiung CA, Wu CW, Wang LH, Chang IS. Upregulation of SOX9 in lung adenocarcinoma and its involvement in the regulation of cell growth and tumorigenicity. Clin Cancer Res. 2010 Sep 1;16(17):4363-73. doi: 10.1158/1078-0432.CCR-10-0138. Epub 2010 Jul 22. PMID 20651055
- [Background] Harley VR, Clarkson MJ, Argentaro A. The molecular action and regulation of the testis-determining factors, SRY (sex-determining region on the Y chromosome) and SOX9 [SRY-related high-mobility group (HMG) box 9]. Endocr Rev. 2003 Aug;24(4):466-87. doi: 10.1210/er.2002-0025. PMID 12920151